CLINICAL TRIAL: NCT07235774
Title: A Phase 1, Open-label, Single-sequence, 2-period Study to Determine the Effects of Repeated Oral Dosing of Vorasidenib on the Pharmacokinetics, Safety and Tolerability of a Combined Oral Contraceptive in Healthy Female Participants.
Brief Title: A Drug-drug Interaction Study of Vorasidenib and a Combined Oral Contraceptive in Healthy Female Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (I.R.I.S.) (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: S095032-234
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Healthy Adult Female Participants
MeSH Terms: interventions — vorasidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vorasidenib and drospirenone (DRSP)/ethinyl estradiol (EE) (Experimental): Participants will receive a single oral dose of 3 mg DRSP/0.02 mg EE on Day 1.
  Participants will receive an oral daily dose of 40mg vorasidenib from Day 6 to Day 24. In addition, participants will receive a single oral dose of 3 mg DRSP/0.02 mg EE on Day 20, co-administered with vorasidenib.
  Interventions: Drug: Vorasidenib; Drug: DRSP/EE

INTERVENTIONS:
Drug: Vorasidenib — 40mg taken orally daily from Day 6 through Day 24
Drug: DRSP/EE — 3 mg DRSP/0.02 mg EE taken orally on Day 1 and Day 20

SUMMARY:
The objective of this study is to evaluate the effect of multiple oral doses of vorasidenib on the single dose pharmacokinetics of the representative combined oral contraceptive, drospirenone (DRSP)/ethinyl estradiol (EE), in healthy female participants. The study includes a screening phase, two treatment periods in-house, and a follow-up period. During the first period, from Day 1 through Day 5, participants will take one dose of DRSP/EE. In the second treatment period, from Day 6 through Day 24, participants will take vorasidenib every day, and on Day 20, they will take DRSP/EE along with vorasidenib. The entire study, including screening and follow-up, will last up to 83 days. Participants may undergo blood tests, heart tests (electrocardiogram (ECG)), vital sign checks, and physical exams.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, nonpregnant, nonlactating pre- or post-menopausal female participants, including women of childbearing potential (WOCBP), assigned female at birth only.
* 18 - 55 years of age (both inclusive) at Screening.
* Body mass index (BMI) of 18.0 - 30.0 kg/m² (both inclusive) at Screening.
* Body weight of at least 40 kg at Screening.
* Participants of childbearing potential who must use two effective methods of birth control (e.g., non-hormonal intrauterine device [IUD], male or female condom with spermicide, cap, diaphragm, or sponge with spermicide), or abstinence, from Screening until at least 90 days after the last dose of vorasidenib or who must be surgically sterile (e.g., hysteroscopic sterilization, bilateral tubal salpingectomy, hysterectomy, or bilateral oophorectomy) at least 6 months prior to the first dose of IMP in the study. Participants of childbearing potential must have a negative serum pregnancy test at Screening and prior to the first dose of IMP in the study.
* Post-menopausal participants (defined as amenorrhea for 12 consecutive months and documented plasma follicle stimulating hormone [FSH] level > 40 IU/mL) who must have a FSH test confirming the post-menopausal status at Screening.
* A continuous nonsmoker who has not used nicotine-containing products (e.g., snuff, nicotine patch, nicotine chewing gum, mock cigarettes, or inhalers) for at least 3 months prior to the first dose of IMP in the study based on a cotinine test result.
* Participants who are considered by the Investigator to be in good general health as determined by medical history, full physical examination, clinical laboratory test results, 12-lead electrocardiogram (ECG) results, and vital sign measurements findings at Screening and Admission.

Exclusion Criteria:

* Participants of childbearing potential who are pregnant, lactating, or planning to become pregnant within at least 90 days after the last dose of vorasidenib; the participants who are on oral contraceptive pills or contraceptive patch within 31 days prior to the first dose of IMP in the study; participants who use a hormonal IUD or vaginal ring within 3 months prior to the first dose of IMP in the study; or participants who receive any injectable or implantable hormone containing product within 1 year prior to the first dose of IMP in the study.
* Participant who consume grapefruit or grapefruit juice, or Seville orange or Seville orange-containing products (e.g., marmalade), within 14 days prior to the first dose of IMP in the study.
* Participant who ingest vegetables from the mustard green family (e.g., kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, and mustard) and charbroiled meats within 14 days prior to the first dose of IMP in the study.
* Participant who consume caffeine- or xanthine-containing products (e.g., coffee, tea, cola drinks, and chocolate), alcohol, or products containing any of these within 48 hours prior to the first dose of IMP in the study.
* Participants who are unable or unwilling to abstain from recreational drugs, alcohol, caffeine, xanthine-containing beverages or food (e.g., coffee, tea, chocolate, and caffeinated sodas, colas), grapefruit, grapefruit juice, Seville oranges, or products containing any of these from 48 hours (caffeine, xanthine-containing beverages or food, alcohol) or 14 days (recreational drugs, grapefruit, grapefruit juice, Seville oranges, or Seville orange-containing products) prior to the first dose of IMP in the study until the Discharge/Early Termination visit.
* In the opinion of the Investigator, participants who are not suitable for entry into the study.
* Participant who have received any vaccine or used any prescription (including hormone replacement therapy) or over-the-counter medications (except acetaminophen/paracetamol [up to 2 g per 24 hours] or ibuprofen [up to 1.2 g per 24 hours]), including herbal (e.g., St. John's Wort) or nutritional supplements, within 14 days or 5 drug half-lives, whichever is longer, prior to the first dose of IMP in the study.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2026-03-14 (Estimated); Study Completion 2026-03-14 (Estimated)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) of DRSP and EE | Through Day 25
Area under the plasma concentration versus time curve (AUC) from time 0 to the last quantifiable concentration (AUC0-last) of DRSP and EE | Through Day 25
AUC from 0 extrapolated to infinity (AUC0-inf) of DRSP and EE | Through Day 25
Time corresponding to Cmax (Tmax) of DRSP and EE | Through Day 25
Terminal half-life (t1/2) of DRSP and EE | Through Day 25
Apparent oral clearance (CL/F) of DRSP and EE | Through Day 25
Apparent volume of distribution during the terminal phase following oral administration (Vz/F) of DRSP and EE | Through Day 25
Elimination rate constant (Kel) of DRSP and EE | Through Day 25

SECONDARY OUTCOMES:
Number of Adverse Events (AEs) | Through the Follow-up Phone Call (Day 53)
Trough plasma concentration (Ctrough) of vorasidenib | Through Day 24

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Belfast, Northern Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorization in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.